CLINICAL TRIAL: NCT01412021
Title: Humira® for Subcutaneous Injection Special Investigation ( All-case Survey ) in Patients With Juvenile Idiopathic Arthritis Study
Brief Title: Special Investigation (All Case Survey) in Patients With Juvenile Idiopathic Arthritis
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P12-769
Record Dates: First submitted 2011-08-05; First posted 2011-08-08 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-01

CONDITIONS: Arthritis, Juvenile Rheumatoid
Keywords: Arthritis, Juvenile Rheumatoid
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Humira: Participants with juvenile idiopathic arthritis who received Humira (adalimumab).

SUMMARY:
This study of Humira will be conducted to clarify the following with regard to the treatment of juvenile idiopathic arthritis affecting multiple joints with this drug:

* Unknown adverse drug reactions (especially important adverse drug reactions)
* Incidence and conditions of occurrence of adverse reactions in the clinical setting
* Factors that may affect the safety and effectiveness of Humira

ELIGIBILITY:
Inclusion Criteria:

* All patients with Juvenile idiopathic arthritis who are not responding well to conventional therapy and receive Humira will be enrolled in the survey

Exclusion Criteria:

* Contraindications according to the Package Insert
* Patients who have serious infections
* Patients who have tuberculosis
* Patients with a history of hypersensitivity to any ingredient of Humira
* Patients who have demyelinating disease or with a history of demyelinating disease
* Patients who have congestive cardiac failure

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who receive Humira for the treatment of Juvenile idiopathic arthritis
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2018-04-02 (Actual); Study Completion 2018-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Package Insert Information — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Humira
Started (registered participants) | 375
Case Report Forms Locked | 368
Completed (Safety Analysis) | 356
Not Completed | 19
Not completed — Case Report Forms Not Retrieved | 7
Not completed — Treatment Prior to Approval | 3
Not completed — Transferred to Other Hospital | 9

BASELINE CHARACTERISTICS:
Population: safety analysis set
Arm/Group | Humira
Number analyzed (Participants) | 356
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241
  Male | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 352
  Other, Not Specified | 4
Disease Activity Scale 28 (DAS28)-4/Erythrocyte Sedimentation Rate (ESR) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 is a validated index of arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, ESR, and the Subject's Global Assessment of Disease Activity (subject rates disease activity using a Likert scale from 0 [low activity] to 10 [high activity]) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission. Population: participants in the efficacy analysis set with an assessment
  units on a scale
    number analyzed (Participants) | 170
    (all) | 3.70 (1.48)
DAS28-4/C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 is a validated index of arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, CRP, and the Subject's Global Assessment of Disease Activity (subject rates disease activity using a Likert scale from 0 [low activity] to 10 [high activity]) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission. Population: participants in the efficacy analysis set with an assessment
  units on a scale
    number analyzed (Participants) | 175
    (all) | 3.42 (1.32)
Serum Matrix Metalloprotease-3 (MMP3) Level [Mean (Standard Deviation); unit: ng/mL] — Population: participants in the efficacy analysis set with an assessment
  ng/mL
    number analyzed (Participants) | 180
    (all) | 162.68 (191.30)
Physician Global Assessment Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: mm] — A VAS was used for the Physician Global Assessment of disease activity (current status). The left end of the VAS scale (0 mm) signifies the absence of symptoms and the right end (100 mm) signifies maximum disease activity. Population: participants in the efficacy analysis set with an assessment
  mm
    number analyzed (Participants) | 169
    (all) | 40.6 (25.1)
Anti-Cyclic Citullinated Peptide Antibody [Mean (Standard Deviation); unit: U/mL] — Population: participants in the efficacy analysis set with an assessment
  U/mL
    number analyzed (Participants) | 115
    (all) | 89.41 (158.34)
Height [Mean (Standard Deviation); unit: cm] — Population: participants in the safety analysis set with an assessment
  cm
    number analyzed (Participants) | 291
    (all) | 143.86 (19.24)
Weight [Mean (Standard Deviation); unit: kg] — Population: participants in the safety analysis set with an assessment
  kg
    number analyzed (Participants) | 299
    (all) | 40.54 (14.51)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in DAS28-4/ESR at Week 4
Description: The DAS28 is a validated index of arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, ESR, and the Subject's Global Assessment of Disease Activity (subject rates disease activity using a Likert scale from 0 [low activity] to 10 [high activity]) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Baseline, Week 4
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 145
units on a scale | -1.01 (1.08)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test; redundancy is not taken into consideration

2. Primary Outcome: Change From Baseline in DAS28-4/ESR at Week 8
Description: as for outcome 1
Time Frame: Baseline, Week 8
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 123
units on a scale | -1.39 (1.26)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test; redundancy is not taken into consideration

3. Primary Outcome: Change From Baseline in DAS28-4/ESR at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 127
units on a scale | -1.39 (1.28)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test; redundancy is not taken into consideration

4. Primary Outcome: Change From Baseline in DAS28-4/ESR at Week 16
Description: as for outcome 1
Time Frame: Baseline, Week 16
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 134
units on a scale | -1.46 (1.40)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test; redundancy is not taken into consideration

5. Primary Outcome: Change From Baseline in DAS28-4/ESR at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 128
units on a scale | -1.64 (1.52)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test; redundancy is not taken into consideration

6. Primary Outcome: Change From Baseline in DAS28-4/CRP at Week 4
Description: The DAS28 is a validated index of arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, CRP, and the Subject's Global Assessment of Disease Activity (subject rates disease activity using a Likert scale from 0 [low activity] to 10 [high activity]) are included in the DAS28 score. Scores on the DAS28 range from 0 to 10. A DAS28 score >5.1 indicates high disease activity, a DAS28 score <3.2 indicates low disease activity, and a DAS28 score <2.6 indicates clinical remission.
Time Frame: Baseline, Week 4
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 155
units on a scale | -0.94 (1.01)

7. Primary Outcome: Change From Baseline in DAS28-4/CRP at Week 8
Description: as for outcome 6
Time Frame: Baseline, Week 8
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 130
units on a scale | -1.24 (1.14)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test; redundancy is not taken into consideration

8. Primary Outcome: Change From Baseline in DAS28-4/CRP at Week 12
Description: as for outcome 6
Time Frame: Baseline, Week 12
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 135
units on a scale | -1.29 (1.12)

9. Primary Outcome: Change From Baseline in DAS28-4/CRP at Week 16
Description: as for outcome 6
Time Frame: Baseline, Week 16
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 140
units on a scale | -1.35 (1.23)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test; redundancy is not taken into consideration

10. Primary Outcome: Change From Baseline in DAS28-4/CRP at Week 24
Description: as for outcome 6
Time Frame: Baseline, Week 24
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Humira
Number analyzed (Participants) | 135
units on a scale | -1.57 (1.36)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test; redundancy is not taken into consideration

11. Primary Outcome: Change From Baseline in Serum MMP3 Level at Week 4
Time Frame: Baseline, Week 4
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Humira
Number analyzed (Participants) | 158
ng/mL | -72.18 (138.24)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

12. Primary Outcome: Change From Baseline in Serum MMP3 Level at Week 8
Time Frame: Baseline, Week 8
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Humira
Number analyzed (Participants) | 131
ng/mL | -83.36 (159.27)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

13. Primary Outcome: Change From Baseline in Serum MMP3 Level at Week 12
Time Frame: Baseline, Week 12
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Humira
Number analyzed (Participants) | 140
ng/mL | -78.05 (144.73)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

14. Primary Outcome: Change From Baseline in Serum MMP3 Level at Week 16
Time Frame: Baseline, Week 16
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Humira
Number analyzed (Participants) | 148
ng/mL | -86.28 (178.51)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

15. Primary Outcome: Change From Baseline in Serum MMP3 Level at Week 24
Time Frame: Baseline, Week 24
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Humira
Number analyzed (Participants) | 146
ng/mL | -98.67 (185.07)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

16. Primary Outcome: Change From Baseline in Physician Global Assessment (VAS) at Week 4
Description: A VAS was used for the Physician Global Assessment of disease activity (current status). The left end of the VAS scale (0 mm) signifies the absence of symptoms and the right end (100 mm) signifies maximum disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 4
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Humira
Number analyzed (Participants) | 152
mm | -15.5 (20.8)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

17. Primary Outcome: Change From Baseline in Physician Global Assessment (VAS) at Week 8
Description: as for outcome 16
Time Frame: Baseline, Week 8
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Humira
Number analyzed (Participants) | 132
mm | -21.5 (23.7)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

18. Primary Outcome: Change From Baseline in Physician Global Assessment (VAS) at Week 12
Description: as for outcome 16
Time Frame: Baseline, Week 12
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Humira
Number analyzed (Participants) | 132
mm | -21.8 (25.8)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

19. Primary Outcome: Change From Baseline in Physician Global Assessment (VAS) at Week 16
Description: as for outcome 16
Time Frame: Baseline, Week 16
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Humira
Number analyzed (Participants) | 136
mm | -25.3 (24.9)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

20. Primary Outcome: Change From Baseline in Physician Global Assessment (VAS) at Week 24
Description: as for outcome 16
Time Frame: Baseline, Week 24
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Humira
Number analyzed (Participants) | 136
mm | -27.0 (27.9)

21. Primary Outcome: Change From Baseline in Anti-Cyclic Citrullinated Peptide Antibodies at Week 24
Time Frame: Baseline, Week 24
Population: participants in the efficacy analysis set with an assessment
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Humira
Number analyzed (Participants) | 33
U/mL | -45.03 (98.58)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p = 0.0132, paired t-test

22. Primary Outcome: Change From Baseline in Height at Week 4
Time Frame: Baseline, Week 4
Population: participants in the safety analysis set with an assessment
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Humira
Number analyzed (Participants) | 152
cm | 0.24 (0.65)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

23. Primary Outcome: Change From Baseline in Height at Week 8
Time Frame: Baseline, Week 8
Population: participants in the safety analysis set with an assessment
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Humira
Number analyzed (Participants) | 130
cm | 0.59 (0.92)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

24. Primary Outcome: Change From Baseline in Height at Week 12
Time Frame: Baseline, Week 12
Population: participants in the safety analysis set with an assessment
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Humira
Number analyzed (Participants) | 146
cm | 0.88 (0.96)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

25. Primary Outcome: Change From Baseline in Height at Week 16
Time Frame: Baseline, Week 16
Population: participants in the safety analysis set with an assessment
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Humira
Number analyzed (Participants) | 154
cm | 1.25 (1.40)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

26. Primary Outcome: Change From Baseline in Height at Week 24
Time Frame: Baseline, Week 24
Population: participants in the safety analysis set with an assessment
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Humira
Number analyzed (Participants) | 164
cm | 1.60 (1.63)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

27. Primary Outcome: Change From Baseline in Weight at Week 4
Time Frame: Baseline, Week 4
Population: participants in the safety analysis set with an assessment
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Humira
Number analyzed (Participants) | 164
kg | 0.47 (1.22)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

28. Primary Outcome: Change From Baseline in Weight at Week 8
Time Frame: Baseline, Week 8
Population: participants in the safety analysis set with an assessment
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Humira
Number analyzed (Participants) | 139
kg | 0.82 (1.56)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

29. Primary Outcome: Change From Baseline in Weight at Week 12
Time Frame: Baseline, Week 12
Population: participants in the safety analysis set with an assessment
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Humira
Number analyzed (Participants) | 158
kg | 1.10 (1.90)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

30. Primary Outcome: Change From Baseline in Weight at Week 16
Time Frame: Baseline, Week 16
Population: participants in the safety analysis set with an assessment
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Humira
Number analyzed (Participants) | 166
kg | 1.37 (2.14)
Statistical Analysis 1: Comparison: Humira; Test type: Superiority; p < 0.0001, paired t-test

31. Primary Outcome: Change From Baseline in Weight at Week 24
Time Frame: Baseline, Week 24
Population: participants in the safety analysis set with an assessment
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Humira
Number analyzed (Participants) | 174
kg | 1.76 (2.34)

32. Other Pre Specified Outcome: Number of Participants With Adverse Drug Reactions (ADRs)
Description: Adverse drug reactions are defined and totaled as collected adverse events whose causal relation with adalimumab cannot be ruled out. An adverse event refers to any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease associated with the use of a drug, whether or not considered related to the drug.
Time Frame: up to Week 24
Population: participants in the safety analysis set with an assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Humira
Number analyzed (Participants) | 356
Participants
  ADRs | 106
  Serious ADRs | 12

ADVERSE EVENTS:
Time Frame: up to Week 24
Arm/Group | Humira
All-Cause Mortality (participants affected / at risk) | 0/356
Serious Adverse Events (participants affected / at risk) | 17/356
Other Adverse Events (participants affected / at risk) | 20/356
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (N=356)
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Disseminated tuberculosis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pulmonary tuberculosis (Infections and infestations) | 1
Salpingitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Water intoxication (Metabolism and nutrition disorders) | 1
Epilepsy (Nervous system disorders) | 1
Febrile convulsion (Nervous system disorders) | 1
Papillophlebitis (Eye disorders) | 1
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Gastric mucosal lesion (Gastrointestinal disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (N=356)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT01412021/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT01412021/SAP_001.pdf